CLINICAL TRIAL: NCT03634930
Title: Josef Ressel Centre for the Investigation of Early Life Metabolic Programming Regarding Dispositions of Obesity
Brief Title: Josef Ressel Centre Perinatal Programming
Acronym: JRP
Status: Recruiting | Type: Observational
Sponsor: Moenie van der Kleyn (Industry)
Collaborators: Christian Doppler Forschungsgesellschaft (Unknown); Milupa GmbH (Industry)
Responsible Party: Sponsor-Investigator, Moenie van der Kleyn, Head of Josef Ressel Centre, FH Joanneum Gesellschaft mbH
Organization: FH Joanneum Gesellschaft mbH (Industry)
Other Study IDs: PJM.16.001.01
Record Dates: First submitted 2018-07-24; First posted 2018-08-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Childhood Obesity
Keywords: Breast Feeding, Exclusive versus Formula Feeding, Exclusive; satiety cues; childhood obesity; biomarker; nutritional status; infant body composition; infant weight gain velocity; metabolic programming; inflammation
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding; Inflammation | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Milk, blood (mother and child), urine (child), saliva (mother and child) and stool sample (mother and child), hair sample (mother and child)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EBF exclusive breast fed children at 16 weeks: observation of 24 hours drinking volume, weight, length, body composition, biomarker and satiety cues, as well as eating- and feeding behaviour and nutritional status of exklusiv breastfed children at the age of 8 and 16 weeks, and at 1 and 2 Years
  Interventions: Behavioral: observation
- EFF exclusive formula fed children at 16 week: observation of 24 hours drinking volume, weight, length, body composition, biomarker and satiety cues, as well as eating- and feeding behaviour and nutritional status of exklusiv formula fed children at the age of 8 and 16 weeks, and at 1 and 2 Years
  Interventions: Behavioral: observation

INTERVENTIONS:
Behavioral: observation — Observation of growth, infant bodycomposition, 24h-drinkingvolume

SUMMARY:
Background: Metabolic imprinting through early childhood nutrition seems to play an important role in the aetiology of obesity. Overweight at age two and later in life is associated with excessive weight gain as early as three months of age. Breastfeeding in the first year of life appears to be protective against obesity development.

Objective: of the "Josef Ressel Centre for Early Life Metabolic Programming of Dispositions of Obesity" is to identify maternal and infant predictors of metabolic risk of obesity. The main considerations of modifiable factors are early infant nutrition, 24-hours-drinking-volume, the velocity of infant weight gain, in relation to infant fat mass and fat free mass, to biomarker and to the nutritional status of the mother. A second focus is put on maternal feeding style, infant eating behaviour and the identification of satiety cues.

Multi-Study design: a monocentric prospective longitudinal cohort of 100 healthy, non-obese, non-smoking pregnant mothers and their term, normal birthweight, singleton babies. Mothers and exclusively breastfed versus exclusively formula fed children (at 16 weeks) will be examined at 36 weeks of pregnancy, 4 - 8 - 12 and 16 weeks of life, follow-up at 1 and 2 years of life.

Methods: four weighing protocols between 4th and 16th week of life, feeding diary, anthropometric data measurement of mother and child, child fat mass index by air displacement plethysmograph. Macronutrient and energy content of the breast milk will be analysed by MIRIS™.

Well-defined biomarkers of oxidative stress and inflammation, lipid profile, adipokines, insulin, as well as micro- und macronutrients will be analysed as meaningful indicators regarding the development of obesity and/or the metabolic syndrome in newborns. Samples, such as plasma, urine, saliva, and stool of the mothers and children will be examined with High Performance Liquid Chromatography, High Performance Gas Chromatography, Mass Spectrometry, Enzyme-Linked Immunosorbent Assay (ELISA) and more. Also questionnaires for the evaluation of the maternal milk feeding style are used as well as the Baby and Child Eating and Behaviour Questionnaire at 16 weeks, 1 and 2 years.

A semi-automatic recognition of infants' satiety cues during feeding will be performed. The recording environment includes video cameras and microphones, a pulse oximeter, etc. All signals are synchronously recorded with the aid of the hardware and software infrastructure.

DETAILED DESCRIPTION:
Nutrition related diseases such as obesity are considered as the main health problems in the 21st century. Overweight and obesity are significant risk factors regarding the development of cardiovascular diseases, strokes, diabetes mellitus, and other non-communicable diseases. In the "Josef Ressel Centre for the Investigation of Early Life Metabolic Programming regarding Dispositions of Obesity" possible predictors towards obesity and their relationship to the volume uptake of formula are to be explored multi-dimensionally. During the first part of the project, the volume study, including a total of 66 mother-infant pairs at the 16th week of life, the overfeeding of infants will be investigated. Overfeeding of infants can be regarded in the context of the amount of food consumed, the ingredients, or in the context of satiety perception of babies by their mother. A closer inspection of the drinking volume of breast-fed infants in comparison to formula-fed ones could give an indication of how much and in what frequency infants ingest food and how the drinking volume affects the weight gain and body fat percentage. To do so, applicable anthropometric data will be collected and the measurement of body fat from mothers and infants will be carried out. Additionally, a semi-automatic detection of satiety signals during feeding will be performed. The identification of satiety signs and the reaction of the mother to those signals, in addition with the feeding style, are related to the weight of the infant and its risk of becoming obese later in life. During the second part of the research project, it will be emphasized whether a coherence exists between early infant nutrition and the manifestation of biomarkers of oxidative stress and inflammation. Thus, detailed analyses regarding macro- and micronutrients, adipokines and biomarkers of oxidative stress of mother milk and biological specimen from mothers and infants will be performed Furthermore, the microbiome of the gut of mothers and infants will be investigated. Results from bioanalytical experiments are intended to sup-port the interpretation of results from the volume study to perceive a deep understanding of the metabolic programming phenomenon of infants at the molecular level.

The five main areas of investigation are:

1. 24-hours-drinking-volume: Background: beyond the quality of nutrition during neonatal life, also the quantity in terms of overfeeding plays a critical role in the development of obesity. Objective: to derive evidence on the drinking volume of exclusively breastfed versus exclusively formula fed children, applying strictly the WHO definitions of exclusivity. Secondary objective is the integration of body composition and growth velocity, which may contribute to insights on critical time slots for programming overweight. Methods: weighing protocol, feeding diary, anthropometric data measurement of mother and child, child fat mass index by air displacement plethysmograph PeaPod™ and BodPod™ of the company Cosmed™. The macronutrient and energy content of the breast milk will be also analyzed by MIRIS™.
2. Nutritional Status of Mother and Child:

   Background: evidence suggests that programming may be induced by even mild intrauterine poor nutrition and may confer an increased risk of obesity, without neonates exhibiting birth weights below or above what is considered to be normal. Objectives: both maternal over- and undernutrition, seen as excess energy intake and/or deficiencies of micro- and macronutrients during (late) pregnancy, may increase infant fat mass. Methods: maternal food frequency questionnaire is adapted for pregnancy, an infant food frequency questionnaire is developed for the time span up to two years.
3. Maternal Feeding Style and Child Eating Behaviour:

   Background: a strong maternal control of eating habits is associated with obesity in childhood. Objectives: a prospective investigation of associations between infant eating behaviour and weight gain to gather evidence on the time of establishment and the causal role of infant eating behaviours in weight gain and BMI at two years. Methods: also questionnaires for the evaluation of the maternal milk feeding style are used as well as the Baby and Child Eating and Behaviour Questionnaire at 16 weeks, 1 and at 2 years.
4. Infant Satiety Cues:

   Background: there is an increasing probability that bottle feeding habits, like encouraging the infants to drink the whole content of the bottle, develops overfeeding habits and causes a lower feeling of satiety. Objective: the identification of satiety cues may directly contribute to an objective method to assess satiety. Methods: a semi-automatic recognition of infants' satiety cues during feeding will be performed. The recording environment includes video cameras and microphones, a pulse oximeter, etc. All signals are synchronously recorded with the aid of the hardware and software infrastructure (Noldus-Observer- XT™, Noldus-Media-Recorder™).
5. Biomarker:

Background and Objectives: well-defined biomarkers of oxidative stress and inflammation, lipid profile, ghrelin, leptin, adipokines insulin, as well as micro- und macronutrients will be analysed as meaningful indicators regarding the development of obesity and/or the metabolic syndrome in newborns. Methods: samples, such as plasma, urine, saliva, and stool of the mothers and children will be examined with High Performance Liquid Chromatography, High Performance Gas Chromatography, Mass Spectrometry, Enzyme-Linked Immunosorbent Assay (ELISA) and more.

.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnancy or mother in puerperium
2. Delivery of baby at 37+0 to 41+6 gestational age
3. Legal age (18 years old), age limit 50 years
4. Written consent of test person after having been informed
5. BMI ≥ 18.5 kg/m² to < 30 kg/m²
6. Negative result of oGTT (oral glucose tolerance test) during pregnancy
7. Birth weight of baby 2.5-4.5 kg
8. Non-smoker since knowledge of pregnancy
9. Very good knowledge of German language and Caucasian
10. Exclusive breastfeeding or exclusive formula feeding at MR 2 (4th week of life)

Exclusion Criteria:

1. Birth before 37+0 week of pregnancy (WoP) or after the 41+6 WoP
2. Multiple pregnancy
3. Children with serious congenital malformations of

   * Nervous system
   * Mouth, throat, neck
   * Circulation system
   * Respiratory tract
   * Gastrointestinal tract
   * Urogenital tract
   * Chromosomal aberrations
4. Diseases or hospitalization or intensive medical care of child during neonatal period
5. Hereditary metabolic diseases of child

   * Hereditary disorders of fat metabolism (MCHAD: Medium Chain Acyl-CoA Dehydrogenase Deficiency, LCHAD: Long Chain Acyl-CoA Dehydrogenase Deficiency, VLCHAD: Very Long Chain Acyl-CoA Dehydrogenase Deficiency)
   * Hereditary disorders of amino acid metabolism (PKU: Phenylketonuria)
   * Hereditary disorders of carbohydrate metabolism (Glycogenosis, Galactosemia, Hereditary fructose intolerance, Diabetes mellitus Type 1)
6. Drug (tobacco) abuse
7. Mental illnesses that have to be treated with medicaments
8. Metabolic or autoimmune diseases of mother
9. Complications at birth (blood loss > 1000 ml or eclampsia)
10. Pre-conceptional diabetes (type 1 or 2)
11. Celiac disease and/or wheat protein allergy of mother
12. Breast surgery and/or hypomastia
13. Mixed feeding at MR 2 (4th week of life)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women and young (breastfeeding) mothers. Babys of both sex
Study Population: term (37-41 gestational age), singleton healthy babies with normal birth weight (2.5-4.5 kg) from healthy, non-smoking, non-diabetic mothers with a normal pre-pregnancy BMI (18.5-30). Pregnant women, who plan to breastfeed will be selected from a primary care clinic (STGKK Graz) and young non-breastfeeding mothers will be selected at the maternity ward of the university hospital of Graz.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in 24 hours drinking volume of milk intake | Changes from 4 to 8 to 12 and to 16 weeks of life
  24 hours drinking volume (milliliter) of milk intake of exclusive breast fed versus exclusive formula fed children by 24h-testweighing on an MBC-15K2DM-Infantscale (Kern).
Changes in Body Mass Index (BMI) child | Changes from 4 to 8 to 12 and to 16 weeks of life up to 1 and 2 years
  weight in kilograms, height in meters will be combined to report BMI in (kg/m^2)
Changes in Fat Mass Index (FMI) child | Changes from 8 to 16 weeks of life and 2 years
  weight of fat mass in kilograms, height in meters will be combined to report Fat Mass Index in kg/m^2). Fat mass will be measured by air displacement plethysmography (ADP) system using whole body densitometry to determine body composition (fat and fat-free mass) using a PEA-POD™ and BOD-POD™ (COSMED Company USA).
Change in energy content of mature breast milk | from 8 to 16 weeks of life
  Change in energy content of 3 ml mature breast milk will be determined by MIRIS HMA™ Human Milk Analyzer (Miris Holding AB, Sweden) in kcal/dL. Samples will be measured twice and mean values for all measured parameters will be calculated. Milk samples are gained by use of Harmony Breast Pump kit (Medela Inc., USA) and are immediately frozen at -80 °C. The samples are collected between 9 and 11 AM from one breast simultaneously to feeding at the other breast. Foremilk and hindmilk are mixed, sample size will be at least 20 ml.
Duration of exclusive milk feeding | over the period from 4 to 8 to 12 and to 16 weeks of life up to 1 and 2 years
  The duration of the exclusivity of human milk- or formula feeding will be determined by means of a prospective feeding diary in which frequency, volume, content, administration form and the initiation of complementary food are recorded by the mother. Precise classification by trained study staff will be according to the WHO categories "sole" (exclusive), "predominant" and "partial" breastfeeding through determination of ratio of total breast milk intake per day to total milk intake of other fluids (like formula milk, water, tea etc.) or foods.

SECONDARY OUTCOMES:
Change of Eating Behaviour - baby | from 8 to 16 weeks of life
  The validated Baby Eating and Behaviour Questionnaire (BEBQ) for parent-reported psychometric measurement of the general appetite of the infant during exclusive milk or formula feeding, containing 18 items measuring 4 appetitive traits: enjoyment of food (EF), food responsiveness (FR), slowness in eating (SE) and satiety responsiveness (SR). All items are scored on a 5-point scale as never, rarely, sometimes, often and always with mean scores for each subscale ranging from 1 to 5. Higher scores indicated higher EF and FR and lower SE and SR.
Change of Eating Behaviour - child | change from 1 year to 2 years of life
  The "Child Eating and behaviour Questionnaire" (CEBQ) is same structured as the BEBQ and is containing 35 items, each rated on a five-point Likert scale that ranges from never to always. Additional to the traits of the BEBQ (Food responsiveness (FR), Enjoyment of food (EF), Satiety responsiveness (SR), Slowness in eating (SE)), four additional scales are added: Emotional over-eating (EOE), Desire to drink (DD), Emotional under-eating (EUE), and Food fussiness (FF). Subscale scores are calculated by taking the mean of the item ratings; higher scores reflect more the behaviour in question.
Change in Maternal Milk Feeding Style - Infant | from 8 to 16 weeks of life
  Infant Milk Feeding Questionnaire (IMFQ) is a standardised multidimensional questionnaire for (self-)assessment of maternal control on food intake and eating habits of the infant (= maternal feeding style). It contains 25 items for measuring maternal control behaviour in 6 categories: 1) encouraging feeding, 2) feeding to a routine, 3) limiting intake, 4) concern for weight, 5) monitoring, 6) perceived responsibility. Each item is on a five-point Likert scale that ranges from never to always or disagree, slightly disagree, neutral, slightly agree, agree. This Questionnaire was modeled on the Child Feeding Questionnaire
Change in Maternal Feeding Style - Child | From 1 year to 2 years of life
  The Child Feeding Questionnaire (CFQ) is a standardised multidimensional questionnaire for (self-)assessment of maternal control on food intake and eating habits of the infant, with a focus on obesity proneness in children. It contains 31 items that can be classified in 7 subscales: 3 subscales that measured aspects of parental control over feeding and 4 that measured specific eating attitudes, perceived responsibility for feeding, and perceived parent weight. Responses to all items were coded on a Likert-type scale ranging from 1 (never/ in disagreement) to 5 (always/in agreement). Higher scores reflect more the behaviour in question.
Changes in dietary intake - maternal | from 36 week of pregnancy to 16 weeks, to 1 year to 2 years of life
  assessed with the "Food frequency questionnaire", a semi-quantitative, self-reported online-questionnaire, realised with the aid of a web-based open-source software
Change in dietary intake - infant | change from 1 year to 2 years of life
  assessed with the "Infant food frequency questionnaire", a semi-quantitative, online-questionnaire, reported by the mother, realised with the aid of a web-based open-source software

OTHER OUTCOMES:
Infant satiety cues of breast- and formula fed children | at 8 weeks of life
  In order to identify satiety cues (as for example swallowing, sucking, relaxation, release of nipple) four video and two audio streams together with the physiological signals (Respiration frequency, Muscle activity (by electromyography) and Pulse and oxygen saturation) will be synchronously recorded with the aid of the IT infrastructure (Noldus-Observer-XT™, Noldus-Media-Recorder™, BIOPAC™ and NONIN-Biosignal-Amplifier-Systems™). The coding of the data will be performed offline by means of manual coding by at least two trained individuals. The classification of events that are required to detect satiety cues (sucking rhythm, sucking breaks, duration, etc.) is based on a coding scheme to be defined. Also analysing body movements based on BAP™ (Body Action and Posture Coding System; Dael, Mortillaro & Scherer, 2012) will be used to categorize breast and bottle fed infants' behaviour. The conformity of the coders will be reviewed by Cohen's Kappa.
Changes in fecal microbial profile | Changes from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  DNA is extracted from both maternal and infant stool samples using the Magnapure Bacterial DNA Kit following the recommended procedures on a Hamilton Starlet workstation. DNA concentration is measured by Picogreen fluorescence. Analysis of fecal microbial profile using 16s rRNA sequencing.
Changes in eicosanoids profiles | Change from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  Oxidative stress biomarker like Eicosanoids, 8-hydroxy-2-deoxy guanosine (8-OH-dG) will be measured by high pressure liquid chromatography-mass spectrometry (HPLC-MS) in maternal plasma, breast milk and urine as well as in infant plasma and urine. Concentration of carbonyl proteins in breast milk and in plasma of mothers and infants will be determiated by enzyme-linked immunosorbent assay (ELISA).
Changes in satiety hormones profiles | Change from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  Concentrations of Leptin, Ghrelin and Irisin will be determined using enzyme-linked immunosorbent assay (ELISA) in breast milk, maternal and infant serum. Salvia samples of mothers and infants will be subjected to cortisol quantification using enzyme-linked immunosorbent assay (ELISA).
Changes in hormone profiles | Change from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  The changes in hormone profiles will be monitored by measuring (Thyroid-stimulating hormone (TSH), triiodothyronine (T3) thyroxine (T4) furthermore Dehydroepiandrosterone sulfate (DHEA-S), Insulin and C-peptide using enzymeimmunoassyay (EIA) by Abbott Architect i2000SR.
Changes in C-reactive protein | Change from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  Biomarker of inflammation will be examinated by measuring C-reactive protein (CRP) in serum or plasma using photometrics on Cobas-c111 (Roche).
Changes in the trace elements levels | Change from 36 week of pregnancy to 8, 16 weeks of life, to 1 and 2 years
  Changes in the trace elements levels (e.g. zinc, selenium, iodine) in maternal plasma and breast milk and in infant plasma will be determinated by tandem mass spectrometry (ICP-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Moenie van der Kleyn, MPH, Study Director — FH Joanneum Hebammen
Locations (1):
- FH Joanneum, university of applied sciences, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Homepage of Josef Ressel Centre for the Investigation of Early Live Metabolic Programming regarding Dispositions of Obesity — https://www.fh-joanneum.at/en/research/josef-ressel-centre-for-research-into-predisposition-to-perinatal-metabolic-programming-of-obesity/
- See also: Homepage of FH Joanneum, university of applied sciences — https://www.fh-joanneum.at/en/